CLINICAL TRIAL: NCT01473992
Title: Comparative Outcomes Assessment of the C-Leg With a New Knee Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Highsmith (Other)
Collaborators: Otto Bock Healthcare (Industry); Florida High Tech Corridor Council (Other)
Responsible Party: Sponsor-Investigator, Jason Highsmith, Principal Investigator, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6140101200
Record Dates: First submitted 2011-05-31; First posted 2011-11-17 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Other and Unspecified Complications of Amputation Stump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prosthetic knee 1 (Otto Bock C-Leg) (Active Comparator): This arm included unilateral transfemoral amputees who were assessed while using their preferred knee at study start(C-Leg). The Otto Bock C-Leg is a microprocessor knee using 2 sensors (1 for kinetics and 1 for kinematics).
  Interventions: Device: Otto Bock C-Leg
- Prosthetic knee 2 (Otto Bock Genium) (Active Comparator): This arm included unilateral transfemoral amputees who were assessed while using the experimental/study knee, the Genium. The Otto Bock Genium is a microprocessor knee using multiple sensors that hypothetically increase mobility functions (e.g. walking backwards, intuitive stance)
  Interventions: Device: Otto Bock Genium
- Non-amputee controls (No Intervention): This was an observational arm including non-amputees who were assessed as non-impaired control subjects. There are no interventions in this observational arm of the study.

INTERVENTIONS:
Device: Otto Bock C-Leg — Amputees' preferred prosthetic knee.
  Arms: Prosthetic knee 1 (Otto Bock C-Leg)
Device: Otto Bock Genium — Study knee.
  Arms: Prosthetic knee 2 (Otto Bock Genium)

SUMMARY:
The purpose of this study is to determine if transfemoral amputees of varied etiology will demonstrate increased function, safety and quality of life following accommodation with a new knee prosthesis as compared to their former C-Leg knee prosthesis.

ELIGIBILITY:
Inclusion criteria:

* Unilateral transfemoral or knee-disarticulation amputee
* 18 to 85 years of age
* K3 (variable cadence and community) ambulators;
* Current use of and experience with the C-Leg for at least 1 year
* Ability to descend stairs and hills without caregiver and assistive devices
* Be able to independently provide informed consent
* Be willing to comply with study procedures.

Exclusion criteria:

* History of chronic skin breakdown on the residual limb
* Conditions that would prevent participation and pose increased risk (e.g. unstable cardiovascular conditions that preclude physical activity such as walking)
* Use of any assistive devices/walking aids, beyond a prosthesis, to ambulate
* Unwillingness/inability to follow instructions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Jason Highsmith, PT,DPT,CP, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prosthetic Knee 1 Then Prosthetic Knee 2: Otto Bock C-Leg: Amputees' preferred prosthetic knee then experimental knee (Genium).
- Prosthetic Knee 2 Then Prosthetic Knee 1: Experimental knee (Otto Bock Genium: Study knee) then subjects' preferred knee (C-Leg).
- Control (Non-amputees): Non-amputee control group
Period: Overall Study
Arm/Group | Prosthetic Knee 1 Then Prosthetic Knee 2 | Prosthetic Knee 2 Then Prosthetic Knee 1 | Control (Non-amputees)
Started | 10 | 10 | 5
Completed | 10 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Otto Bock C-Leg (prosthetic knee 1), amputees' preferred prosthetic knee, first and Otto Bock Genium (prosthetic knee 2), the study knee, first.
- Non Amputee Control Group: non-amputee healty controls
- Total: Total of all reporting groups
Arm/Group | Entire Study Population | Non Amputee Control Group | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (14.2) | 57.2 (15.7) | 51.9 (15.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 3 | 21
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 16 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: 75 Meter Self Selected Walking Test
Description: Time to Complete a 75 meter walking distance.
Time Frame: Based on preliminary experience with the intervention, accommodation can range from 2 weeks to 3 months. Assessment will be scheduled within 2 weeks following accommodation.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Prosthetic Knee 1: Otto Bock C-Leg: Amputees' preferred prosthetic knee.
- Prosthetic Knee 2: Otto Bock Genium: Study knee.
- Non Amputee Control Group: healthy, non-amputee controls
Arm/Group | Prosthetic Knee 1 | Prosthetic Knee 2 | Non Amputee Control Group
Number analyzed (Participants) | 20 | 20 | 5
seconds | 65.1 (10.2) | 64.0 (10.3) | 54.0 (6.9)

2. Secondary Outcome: Balance and Stability
Description: Balance and stability will be assessed for limits of stability using the Biodex SD. The limit of stability score is a scaled score with a possible range of 0 (worst possible outcome) to 100 (best possible outcome)based on variability of the trajectory of the center of mass while weight shifting on a force platform.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prosthetic Knee 1 | Prosthetic Knee 2 | Non Amputee Control Group
Number analyzed (Participants) | 10 | 10 | 5
scores on a scale | 60.7 (24.3) | 59.2 (25.4) | 73.1 (21.3)

3. Secondary Outcome: Prosthesis Evaluation Questionnaire: Utility Score.
Description: The Prosthetics Evaluation Questionnaire (PEQ) was used as a validated survey to solicit participants' subjective experience and feedback regarding prosthesis-related function and quality of life. PEQ domains are ordinally scaled from 0 (worst or most negative feeling/response) to 7 (best or most positive feeling/response).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Prosthetic Knee 1 | Prosthetic Knee 2
Number analyzed (Participants) | 20 | 20
score on a scale | 6.0 [2 to 7] | 5.5 [2 to 7]

4. Primary Outcome: Physical Functional Performance (Continuous Scale; 10-items)
Description: Simulation of 10 activities of daily living (i.e. donning a shirt, sweeping, walking stairs). Measured in units of time, distance and mass to provide a singular, continuous scaled score of function (from 0-100). A score of 100 is the maximal score and indicates the highest level of independent function where a score of 0 indicates the poorest score. Persons scoring lower scores will likely be at increased risk of dependency with daily function.
Time Frame: Accommodation with knee systems is approximately 90 days. This test takes less than 1hr to complete.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Non Amputee Control Group: healthy, non-amputee control group
Arm/Group | Prosthetic Knee 1 | Prosthetic Knee 2 | Non Amputee Control Group
Number analyzed (Participants) | 20 | 20 | 5
scores on a scale | 55.2 (14.8) | 59.6 (16.0) | 73.04 (15.67)

ADVERSE EVENTS:
Arm/Group | Prosthetic Knee 1 | Prosthetic Knee 2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No